CLINICAL TRIAL: NCT05055206
Title: A Feasibility Trial of Lymphatic Mapping With SPECT-CT for Evaluating Contralateral Disease in Lateralized Oropharynx Cancer Using 99m-Technetium Sulfur Colloid
Brief Title: Study of Lymphatic Drainage Mapping in Oropharyngeal Cancers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SPECT-CT; 20-5607 (Other: UHN)
Record Dates: First submitted 2021-09-14; First posted 2021-09-24 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Oropharynx Cancer
Keywords: Lymphatic Drainage Mapping; 99m-Technetium Sulfur Colloid
MeSH Terms: conditions — Oropharyngeal Neoplasms | interventions — Single Photon Emission Computed Tomography Computed Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lymphatic drainage mapping in patients with oropharynx cancer (Experimental): Participants will be given 4 to 6 injections of the radiotracer 99m-Technetium Sulfur Colloid by a needle into one of the veins of the radiotracer around the tumour.
  Participants will then have at least 1 or possibly 2 SPECT-CT scans (a special x-ray scan of the body from many angles that are turned into 3-dimensional pictures on a screen).
  Interventions: Diagnostic Test: SPECT-CT

INTERVENTIONS:
Diagnostic Test: SPECT-CT — 99m-Technetium Sulfur Colloid will be injected prior to the scan.

SUMMARY:
The purpose of the study is to see how practical it is to inject a radiotracer called 99m-Technetium Sulfur Colloid around the tumors for the imaging of patients with oropharyngeal cancer.

DETAILED DESCRIPTION:
This study will evaluate a technique called lymphatic drainage mapping. This is a technique where a radiotracer (a radioactive material that can be seen with a special computed tomography [CT] scanner to create 3D images) is injected into a vein around the tumour, either with local anesthesia or under general anesthesia. The radiotracer that will be used for the lymphatic drainage mapping is called 99m-Technetium Sulfur Colloid. Images will be taken of neck to detect the movement of the radiotracer. This will allow the doctors to see the drainage pattern of the lymph nodes in the neck.

The information from this study will be used to better understand the tendency for oropharyngeal cancers to spread to lymph nodes. In addition, the information from this clinical trial will be used in future clinical studies to help specialists identify strategies to help plan treatment based on this type of imaging study.

ELIGIBILITY:
Inclusion Criteria:

* Patient has lateralized oropharyngeal carcinoma (tonsil or tongue base) not involving midline
* Has squamous cell carcinoma, T1-3 tumours, with no contralateral nodes on clinical exam or axial imaging
* Human papillomavirus (HPV) positive or negative
* Patient should have normal organ function as per Investigator judgement
* Patient is planned for definitive or adjuvant radiotherapy (RT) or chemo radiotherapy (CRT) with bilateral neck RT, or surgery
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1

Exclusion Criteria:

* T4 tumours
* Contralateral/bilateral nodal disease or node(s) > 6cm on clinical exam or axial imaging or positron emission tomography (PET)
* Primary tumour involving or crossing midline
* Soft palate or posterior pharyngeal wall tumour subsites
* Previous head and neck cancer
* Previous radiotherapy (RT) to the head and neck
* Previous neck dissection
* Distant metastases
* Prior invasive malignancy (except non-melanoma skin cancer) unless disease free for 3 years
* Prior radiotracer allergy
* Multiple primary head and neck cancers
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-09-13 (Actual); Primary Completion 2023-10-23 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Proportion of patients injected with radiotracer. | 1 year
Proportion of patients requiring general anesthetic over local anesthetic. | 1 year
Proportion of patients with images that failed radiotracer migration to either side of the neck. | 1 year
Proportion of patients completing 30 minute scan. | 1 year
Proportion of patients completing 3 hour scan. | 1 year
Proportion of patients with radiotracer uptake into a radiographically positive lymph node. | 1 year
Proportion of patients with injections site locations that are compliant with protocol specific map of injection locations. | 1 year
Average time from start to finish of injection of procedure. | 1 year
Proportion of patients with complications associated with injection. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: John de Almeida, M.D., Principal Investigator — University Health Network, Toronto
Locations (4):
- Canada (4):
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No